CLINICAL TRIAL: NCT00936143
Title: An Open Trial to Evaluate the Efficacy and Safety of Infliximab(Remicade) in Treating Patients With Early Ankylosing Spondylitis
Brief Title: Efficacy and Safety Study of Infliximab (Remicade) to Treat Early Ankylosing Spondylitis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Gu Jieruo (Other)
Responsible Party: Sponsor-Investigator, Gu Jieruo, Rheumatology Department, Third Affiliated Hospital of Sun Yat-sen University, Sun Yat-sen University
Organization: Sun Yat-sen University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: REM-CHN-IIS-01
Record Dates: First submitted 2009-07-07; First posted 2009-07-09 (Estimated); Last update posted 2016-01-26 (Estimated); Status verified 2016-01

CONDITIONS: Spondylitis
Keywords: Spondylitis, Ankylosing; infliximab; Antibodies, Monoclonal
MeSH Terms: conditions — Spondylitis; Spondylitis, Ankylosing | interventions — Infliximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- infliximab (Experimental): 200mg infliximab inject intra-venous on baseline, 2nd week, 6th week, 12th week, 24th week
  Interventions: Drug: infliximab

INTERVENTIONS:
Drug: infliximab — 100mg/bottle 5mg/kg inject intra-venous on baseline, 2nd week, 6th week, 12th week, 24th week
  Other Names: remicade

SUMMARY:
This is a prospective open-label study to evaluated the efficacy and safety of infliximab(Remicade) in treating of patients with early ankylosing spondylitis (AS). Infliximab was injected intra-venous on baseline, 2nd week, 6th week, 12th week and 24th week, with dosing of 5mg/kg. The major outcome index is ASAS20, and minor outcome indexes include ASAS50 and ASAS70, BASDAI20,BASDAI50 and BASDAI70. And MRI of sacroiliac joint is not necessary. The adverse events at any time were recorded.

ELIGIBILITY:
Inclusion Criteria:

1. 16 to 65 years old, having signed the informed consent;
2. fulfill the ESSG criteria for diagnosis of SpA; not fulfill the 1984 modified NewYork criteria for AS;
3. have inflammatory back pain defined by Calin criteria;
4. disease duration range from 6 months to 2 years;
5. BASDAI score more than 4;
6. MRI score of sacroiliac joint more than 4;
7. lab examination: hemoglobin more than 90 gram/liter. Aspartate aminotransferase and Alanine aminotransferase less than 2 fold of upper level of normal range. Creatine less than upper level of normal range.

Exclusion Criteria:

1. History of psoriasis or inflammatory bowel disease.
2. Intra-articular injection of cortisone within 3 months.
3. Patients were taking cortisone, SASP or MTX, unless the dose has been stable for at least 3 months.
4. Active iritis.
5. History of heart failure, multiple sclerosis, COPD, lymphoma or other tumor, tuberculosis.
6. Female of pregnancy or breast feeding.
7. History of mental disease and poor compliance.
8. History of drug abuse or alcoholism.

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2008-01; Primary Completion 2009-09 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Proportion of patients achieving ASAS20 improvement. | 6th week

SECONDARY OUTCOMES:
Proportion of patients achieving ASAS50 and ASAS70 | 6th week and 24 week.

CONTACTS AND LOCATIONS:
Locations (1):
- Third Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong, China